CLINICAL TRIAL: NCT06735443
Title: Comparison Of Dexmedetomidine Versus Tramadol As An Adjuvant With Bupivacaine In Caudal Block For Intra-Operative Hemodynamic Stability And Post-Operative Pain In Children Undergoing Inguinal Hernia Surgery
Brief Title: Comparative Efficacy & Safety of Dexmedetomidine vs Tramadol in Paeds Hernioraphy. A Caudal Anaesthesia Approach
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sahiwal medical college sahiwal (Other Government)
Collaborators: Department of medical education (Unknown)
Responsible Party: Principal Investigator, Hafiz Dr Naeem Abbas, Resident Anaesthetist, Sahiwal medical college sahiwal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2094/SLMC/SWL
Record Dates: First submitted 2024-12-04; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Hemodynamic Stability; Post Operative Pain; Inguinal Hernia Repair
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Tramadol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bupivacaine with Dexmetedomidine group (Experimental): In group A, patients will be given 0.25% bupivacaine 1 mL/kg with dexmedetomidine 0.5μg/kg
  Interventions: Drug: Bupivacaine with Dexmetedomidine
- Bupivacaine with Tramadol group (Experimental): In group B, patients will be given 0.25% bupivacaine 1 mL/kg with 1 mg/kg of tramadol
  Interventions: Drug: Bupivacaine with Tramadol

INTERVENTIONS:
Drug: Bupivacaine with Dexmetedomidine — children will be anesthetized generally using Propofol 2.5mg/kg bodyweight, Atracurium 0.5mg/kg body weight and appropriately sized endotracheal tube (ETT) according to the age. Patients will be given 0.25% bupivacaine 1 mL/kg with dexmedetomidine 0.5μg/kg. Neostigmine 0.05mg/kg plus Glycopyrrolate 0.2mg/1mg of neostigmine will be used as reversal agents. After surgery, children will be shifted in post-surgical wards and will be followed-up there for 24 hours. After 24hours, children will be assessed for postoperative pain score.
  Other Names: Bupicain with Dex
  Arms: Bupivacaine with Dexmetedomidine group
Drug: Bupivacaine with Tramadol — children will be anesthetized generally using Propofol 2.5mg/kg bodyweight, Atracurium 0.5mg/kg body weight and appropriately sized endotracheal tube (ETT) according to the age. Patients will be given 0.25% bupivacaine 1 mL/kg with 1 mg/kg of tramadol. Neostigmine 0.05mg/kg plus Glycopyrrolate 0.2mg/1mg of neostigmine will be used as reversal agents. After surgery, children will be shifted in post-surgical wards and will be followed-up there for 24 hours. After 24hours, children will be assessed for postoperative pain score.
  Other Names: Bupicain with Tramal
  Arms: Bupivacaine with Tramadol group

SUMMARY:
Among the postoperative adverse effects, pain has significant importance. Caudal block is a common technique for pediatric analgesia for infraumbilical surgeries. Because of the shortduration of analgesia with bupivacaine alone various additive have been used to prolong the action of bupivacaine. Tramadol has a centrally acting analgesic effect via opioid receptors.Adding Dexmedetomidine to bupivacaine has proven effectiveness for postoperative painrelief. But not much research has been conducted before regarding this comparison which can help us to find the more effective drug for induction of anesthesia.So we want to conduct this randomized trial. Sample size of 60 cases; 30 cases in each group will be included through Nonprobability convenience sampling and will be randomly divided in two groups. In group A,patients will be given 0.25% bupivacaine 1 mL/kg with dexmedetomidine0.5 μg/kg. In group B, patients will be given 0.25% bupivacaine 1 mL/kg with 1mg/kg of tramadol. Heart rate and mean arterial pressure will be assessed before induction of anesthesia, after 5, 10, 15 and 30 mins of induction and at the time of extubation. After surgery, total duration from surgery and first rescue analgesia will be noted. All the information will be recorded on proforma. Data will be entered & analyzed by using SPSS version 20. Both groups will be compared for mean heart rate, MAP and time to first rescue analgesia by using independent samples t-test. P-value ≤0.05 will be considered as significant. So this study will be done in a local setting to get local evidence and implement the use of more appropriate drug with less postop complications, especially in pediatric age group patients. This will help to improve our practice and local guidelines.

DETAILED DESCRIPTION:
After taking approval from hospital ethical committee, 60 children fulfilling the selection criteria will be included in the study from ward of Department of Pediatrics, DHQ Teaching Hospital, Sahiwal. An informed consent will be taken. Demographic information (name, age,gender, weight, ASA and duration of surgery) will be noted.Then children will be randomly divided in two groups by using lottery method for caudal block. In both groups children will be anesthetized generally using Propofol 2.5mg/kg bodyweight, Atracurium 0.5mg/kg body with dexmedetomidine 0.5μg/kg. In group B, patients will be given0.25% bupivacaine 1 mL/kg with 1mg/kg of tramadol. All anesthesia procedures will be done by researcher under supervision of senior consultant anesthesiologist having 4 years residency experience. Heart rate and mean arterial pressure will be assessed after 5,10,15 and 30 mins of induction and at the time of extubation.Neostigmine 0.05mg/kg plus Glycopyrolate 0.2mg/1mg of neostigmine will be used as reversal agents. After surgery, children will be shifted in post-surgical wards and will be followed-up there for 24 hours. Children will be assessed for postoperative pain score. If pain score will be greater than or equal to 5 on FLACC scale, then rescue analgesia will be given and total duration from surgery and first rescue analgesia will be noted (as per operational definition). All the information will be recorded on proforma attached.

definition). All the information will be recorded on proforma (attached). pressure will be assessed before induction of anesthesia, after 5, 10, 15 and 30 minutes weight and appropriate sized endotracheal tube (ETT) according to the age. In group A, patients will be given 0.25% bupivacaine 1 mL/kg

ELIGIBILITY:
Inclusion Criteria:

* Children of age 5-15 years.
* Either gender,
* Elective inguinal hernia surgery.
* ASA I-II
* Proposed duration of surgery <60 minutes.

Exclusion Criteria:

* • Emergency surgery

  * Children with evidence of infection at back, allergy to trial drugs, bleeding/coagulation disorder (PT>15sec), history of developmental delay, sepsis, pre-existing neurological or spinal diseases (on medical record)
  * Expected duration of surgery >120 minutes

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-03-06 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Hemodynamic Stability | Heart rate will be assessed before induction of anesthesia, after 5, 10, 15 and 30 minutes of induction and at the time of extubation.
  heart rate
Post Op Analgesia | After 24hours, children will be assessed for postoperative pain score
  post operative first rescue analgesia
Hemodynamic Stability | Blood pressure will be assessed before induction of anesthesia, after 5, 10, 15 and 30 minutes of induction and at the time of extubation.
  Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Adeel Riaz, MD, Study Director — Sahiwal Teaching Hospital, Sahiwal
Locations (1):
- Sahiwal Medical College Sahiwal, Sahiwal, Punjab Province, Pakistan